CLINICAL TRIAL: NCT01750567
Title: A Phase II Pilot Study of Metformin Therapy in Patients With Relapsed Chronic Lymphocytic Leukemia and Untreated CLL Patients With Genomic Deletion 11q
Brief Title: A Pilot Study of Metformin Therapy in Patients With Relapsed Chronic Lymphocytic Leukemia (CLL) and Untreated CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2012.025
Record Dates: First submitted 2012-10-02; First posted 2012-12-17 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Chronic Lymphocytic Leukemia
Keywords: Relapsed Chronic Lymphocytic Leukemia; untreated CLL patients; genomic deletion 11q
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Metformin (Glucophage) (Experimental): The starting dose of metformin will be 500 mg po daily for one week. The dose can be escalated to 500 mg twice a day after one week, and further escalated to the final dose of 1000 mg twice a day in week 3 if the medication is tolerated without adverse side effects (refer to holding parameters described in section 9.3.3). All doses should be administered with food to decrease gastrointestinal upset.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is an antidiabetic drug which is an inexpensive and generally well tolerated medication.
  Other Names: Glucophage

SUMMARY:
Metformin is an antidiabetic drug which is an inexpensive and generally well tolerated medication. More recently metformin has been shown to act against carcinomas by two mechanisms: 1) an indirect, insulin-dependent mechanism which sensitizes tissues to insulin, inhibits hepatic gluconeogenesis, and stimulates uptake of glucose in muscle, thereby reducing fasting blood glucose and circulating levels of insulin, lowering the pro survival activity of the insulin/INSR axis, and 2) a direct, insulin-independent mechanism which activates the AMP-activated protein kinase (AMPK) pathway and leads to inhibition of the mTOR pathway. Given the investigators preliminary published data on insulin and mTOR inhibition[1] metformin is an attractive candidate for a pilot clinical trial in CLL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have a confirmed diagnosis of chronic lymphocytic leukemia defined as all of the following:

   * ALC > 5000
   * Positive for either CD19 or CD 20 together with CD23 and CD5.
   * Less than 55% atypical cells
2. Patients who relapse after receiving a one or more courses of fludarabine, bendamustine, cytoxan, rituxan, chlorambucil, or campath based therapy.
3. Patients should have findings of relapse by one or both of the following:

   * ALC > 5000 on 2 consecutive occasions and increasing
   * Any increase in lymphadenopathy over best response that has persisted for more than 3 months
4. Patient with confirmed del11q mutation may be included if untreated.
5. Age > or equal to 18 years old and < 80 years of age during the course of therapy
6. ECOG performance 0-2
7. Life expectancy > 12 months
8. Patients must have normal organ function as defined as below:

   * AST and ALT < 2 times the upper limit of normal
   * alkaline phosphatase < 2 ULN
   * serum conjugated bilirubin < 1.5 ULN (exception of Gilbert disease)
   * serum creatinine less than or equal to 1.5 in males, or 1.4 in females
   * GFR > 59
9. Ability to understand and the willingness to sign a written informed consent document
10. Patient must be able to drink and eat more than 75% of their usual daily meals.

Exclusion Criteria:

1. Patients with active CLL disease requiring urgent chemotherapy
2. Patients may not be receiving any other investigational agents.
3. Patients less than 30 days from last treatment for CLL.
4. History of allergic reactions attributed to metformin or other biguanides.
5. Known diabetes (type 1 or 2), fasting glucose > or equal to 7.0 mmol/L (126 mg/dL), or HgbA1C > 6.5
6. Currently taking metformin, sulfonylureas, thiazolidinediones or insulin for any reason
7. Current or planned pregnancy or lactation in women of child bearing age (confirmed by negative pregnancy test prior to start of therapy).
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and sepsis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
9. Conditions which would increase risk of lactic acidosis including:

   * Known alcoholism or ingestion of more than 3 alcoholic beverages per day
   * History of congestive heart failure defined as NYHA class III or IV
   * History of metabolic acidosis
   * Ongoing or active infection concerning for sepsis or SIRS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | Until the patient meets failure criteria and stops Metformin; up to 6 months after start of metformin therapy and yearly thereafter.
  While patients are on metformin therapy, time to treatment failure will be defined as one or all of the following criteria:
  1. ALC > 5000 on 3 occasions after start of metformin treatment and increasing by 25% or more on each occasion, which will be measured every 3 months.
  2. An increase of Rai Stage (0-3) by one stage.
  3. An increase in any lymph node by >50% as assessed by either physical exam (all patients) or CT scanning (only if ordered as part of routine clinical management).
  4. Worsening cytopenias (Hemoglobin <11 g/dl) associated with a bone marrow biopsy result indicating advanced stage CLL (packed CLL marrow).

SECONDARY OUTCOMES:
Time to first therapy (TTFT) in previously untreated 11q CLL subsets only. | from time of diagnosis to time of first treatment with anti-neoplastic chemotherapy.
  To evaluate TTFT in untreated patients, the product-limit method of Kaplan and Meier will be used similarly to the primary endpoint. The main difference between this endpoint and the primary endpoint is that TTFT will be defined from the date of CLL diagnosis for untreated delq11 patients
Changes in the rate of increase of absolute lymphocyte count while on metformin therapy | Until the patient meets failure criteria and stops Metformin
  Longitudinal lymphocyte counts will be modeled using mixed models methodology, whereby both fixed effects (dose of metformin) and random effects (intercept - starting lymphocyte count) can be modeled.
Change in size of clinically appreciated lymphadenopathy in cm and splenomegaly while on metformin therapy | Baseline up to 3 months after completing metformin therapy
  The proportion of patients that begin metformin therapy with these conditions will be summarized, along with the proportions at study defined clinical assessment points during therapy. No statistical models will be employed, but proportions and 95% exact binomial confidence intervals will be reported for descriptive purposes.
Change in number of clinically appreciated lymphadenopathy and splenomegaly while on metformin therapy | Baseline up to 3 months after completing metformin therapy
  The proportion of patients that begin metformin therapy with these conditions will be summarized, along with the proportions at study defined clinical assessment points during therapy. No statistical models will be employed, but proportions and 95% exact binomial confidence intervals will be reported for descriptive purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Sami Malek, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States